CLINICAL TRIAL: NCT03115580
Title: Optical Coherence Tomography Predictors of Functionally Significant Side Branch Compromise After Provisional Main Vessel Stenting In Calcific Coronary Artery Disease Assessed by Fractional Flow Reserve
Brief Title: Side Branch FFR After Provisional Stenting
Acronym: ORBID-FFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Annapoorna Kini, Director Cardiac Cath lab, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-0204
Record Dates: First submitted 2017-04-03; First posted 2017-04-14 (Actual); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Atherectomy, Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Rotational atherectomy (Active Comparator): Rotational atherectomy (RA)
  Interventions: Device: Rotational atherectomy
- CBA/PTCA (Active Comparator): Cutting Balloon Angioplasty (CBA) or Percutaneous transluminal coronary angioplasty (PTCA)
  Interventions: Device: Cutting Balloon Angioplasty

INTERVENTIONS:
Device: Rotational atherectomy — Rotational atherectomy for the treatment of bifurcation lesions to remove plaque with minimal injury to adjacent normal arterial segments and potentially reduce plaque shifting, the "snow plow" effect.
  Other Names: RA
  Arms: Rotational atherectomy
Device: Cutting Balloon Angioplasty — Cutting balloon is a special balloon catheter with three or four microsurgical blades attached longitudinally to its surface, suitable for creating discrete longitudinal incisions in the atherosclerotic target coronary segment during balloon inflation. Lesion preparation will be performed using Cutting Balloon or conventional balloon
  Other Names: CBA
  Arms: CBA/PTCA

SUMMARY:
The purpose of this study is to predict any changes in the side branch after stenting the main branch blood vessel using three dimensional intravascular images. (Frequency domain optical coherence tomography FD OCT).

Optical coherence tomography (OCT) is an established medical imaging technique that uses light to capture high-resolution, three-dimensional images of blood vessels. These images will be used before and after implanting the stent in the main blood vessel. Fractional Flow Reserve (FFR) test, which makes it possible for the interventional cardiologist to calculate blood flow across an area of a coronary artery, will be done after stenting and will help to determine if there are any changes in the side branch blood flow.

DETAILED DESCRIPTION:
Coronary artery bifurcation lesion is a common lesion subset in PCI accounting for 15-20% of the total number of interventions. Treatment of coronary artery bifurcation lesions represents a challenging area in interventional cardiology. When compared with non-bifurcation interventions, bifurcation interventions have a lower rate of procedural success, higher procedural costs, longer hospitalization and a higher clinical and angiographic restenosis. Factors contributing to this adverse outcome include limitations of angiography in assessment of side-branch (SB) disease severity and the lack of established angiographic predictors of SB patency and lumen compromise. Better understanding of the underlying plaque morphology and plaque composition may facilitate more effective treatment of bifurcation lesions.

Intravascular imaging has provided new understanding of mechanisms associated with SB compromise following bifurcation PCI. Plaque shift has been traditionally considered as the principal mechanism for side-branch compromise after main vessel intervention. Rotational atherectomy(RA) has been advocated for the treatment of bifurcation lesions, since it can effectively remove plaque with minimal injury to adjacent normal arterial segments and potentially reduce plaque shifting, the "snow plow" effect. Intravascular ultrasound (IVUS) has been used for guidance in bifurcation lesions, aiding the visualization of plaque morphology at the main vessel and the side-branches and helping the selection of stent size and length as well as the selection of stenting strategy. However, due to the low spatial resolution of IVUS, all attempts for three-dimensional visualization have only focused on visualization of the luminal contour and not on the vessel morphology or the vessel-stent interaction. Optical coherence tomography (OCT) has ~10 times higher resolution than IVUS, which allows precise evaluation of the microstructure of the vessel wall including lipid pool, fibrous cap, calcification, and thrombus. OCT has been shown to constitute a valuable tool for PCI guidance and also the utility of three-dimensional (3D) renderings for assessing the mechanism of side-branch compromise following intervention in bifurcation lesions. The recent development of OCT with online 3D reconstruction allows the operator to obtain a 3D visualization of the lesion and may provide a unique tool for guidance during complex bifurcation PCI and potentially improve stenting results. 3D OCT has been used to visualize jailed side branches after implantation of bioresorbable scaffolds in the main branch and develop a new classification system based on the number of SB compartments. In addition, its potential clinical application in guiding the rewiring of the distal compartment of the SB ostium (jailed with stent struts after MB stenting) to minimize the risk of floating struts was demonstrated It is important to note that while OCT, 3D-OCT, and 3D-QCA (such as that used in the ORBID trial) are imaging modalities that can be used to answer important research questions, their wide-spread adoption in daily clinical practice has been very limited. Intravascular ultrasound (IVUS) is used more frequently as part of a PCI guidance strategy in daily clinical practice.

Fractional flow reserve (FFR) is a pressure-derived, lesion specific index used to determine the functional significance of coronary artery stenosis. Several studies showed that FFR is a safe and feasible method to assess the significance of an ostial SB stenosis after provisional stenting. Quantitative coronary angiography (QCA) has been shown to be unreliable in assessing the functional significance of SB after stent implantation in MV (the area under the curve 0.64, 41.5% sensitivity and 83.1% specificity) suggesting that treatment decisions for jailed SB should not be based on angiographic findings alone. A recent report demonstrated a better ability of post-PCI 3D-OCT to predict the functional significance for SB ostial lesions caused by a jailed SB outcome.

A previous study (ORBID) of 30 patients was done at Mount Sinai Hospital and aimed to identify the predictors of side branch (SB) ostial stenosis developed after provisional stenting of the main vessel (MV) using Optical Coherence Tomography (OCT). The study Showed that High lipid content of the MV lesion and a contralateral location of lipid in the bifurcation area may contribute to SBOS after provisional stenting.

The objective of this study is to analyze the incidence of SB compromise after provisional main vessel stenting in calcified bifurcation lesions of CAD patients, determine the incidence and OCT predictors of functionally significant SB stenosis defined as FFR ≤ 0.8 and to compare the FFR values with 3D-OCT measurements of jailed SB ostium after MV stenting.

Stable CAD patients with bifurcation lesions in whom provisional stenting strategy is planned, who have moderate or severe calcification in the main vessel lesion identified by angiography, SB stenosis 30-70% and SB reference diameter > 2mm will be enrolled in the study.

Moderate calcification will be defined as radiopaque density observed only during the cardiac cycle and typically involving only one side of the vascular wall, and severe calcification will be defined as radiopaque density noted without cardiac motion prior to contrast injection and involving both sides of the arterial wall. After completion of diagnostic angiogram and confirmation of subject eligibility, subjects will be randomly assigned to Rotational Atherectomy (RA) or Cutting Balloon Angioplasty (CBA)/Percutaneous Transluminal Coronary Angioplasty (PTCA) group in a 1:1 fashion.

Patients in both groups will undergo PCI with stent implantation according to current standards of care. Lesion preparation including lesion pre-dilation, scoring or sculpting balloon angioplasty, and use of atherectomy and protection devices will be performed at the operator's discretion, followed by MV stenting. The operator will also decide in both groups about the length and size of the implanted stent. Procedural optimization, such as post-dilation or additional stent implantation will be performed based only on the angiographic findings, according to the discretion of the operator.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age presenting with stable coronary artery disease.
* Patients must have a clinical indication for coronary intervention.
* Creatinine Kinase Myocardial-Band Isoenzyme (CK-MB) must be less than or equal to the upper limit of lab normal (ULN) value within eight hours prior to the procedure.
* The target lesion must be a de novo calcified bifurcation coronary lesion that hasn't been previously treated with any interventional procedure for which provisional main vessel stenting strategy is planned after reviewing angiogram.
* The target vessel must be a native coronary artery with

  1. stenosis ≥70% and <100%, or
  2. Stenosis ≥50% and <70% with evidence of clinical ischemia via positive stress test, or FFR ≤ 0.8, or IVUS or OCT minimal lumen area ≤ 4.0 mm2.
* The target lesion should have SB DS 30 - 70%.
* The target main vessel reference diameter must be ≥2.5 mm and ≤ 4.0 mm.
* The SB reference diameter must be > 2 mm by coronary angiogram.
* The target vessel must have a Thrombolysis in Myocardial Infarction (TIMI) flow grade 3 at baseline.

Exclusion Criteria:

* Patients with ostial left main artery lesions or ostial right coronary artery lesions
* Female patients with child bearing potential not taking adequate contraceptives or currently breastfeeding
* Known allergy to acetylsalicylic acid or clopidogrel.
* Planned surgery within 12 months.
* History of bleeding diathesis
* Major surgery within 15 days
* Life expectancy < 12 months.
* Patients with kidney dysfunction (CrCl<30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annapoorna Kini, MD, MRCO, FACC, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai and the Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between May 2017 and March 2019.
Groups:
- Rotational Atherectomy: Rotational atherectomy (RA) for the treatment of bifurcation lesions to remove plaque with minimal injury to adjacent normal arterial segments and potentially reduce plaque shifting, the "snow plow" effect.
Period: Overall Study
Arm/Group | Rotational Atherectomy | CBA/PTCA
Started | 35 | 36
Completed | 35 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotational Atherectomy | CBA/PTCA | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (10.5) | 66.6 (9.9) | 67.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 21
  Male | 28 | 22 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes Mellitus [Count of Participants; unit: Participants] | 11 | 14 | 25
Hypertension [Count of Participants; unit: Participants] | 28 | 30 | 58
Hyperlipidemia [Count of Participants; unit: Participants] | 32 | 29 | 61
Current smoker [Count of Participants; unit: Participants] | 5 | 1 | 6
Previous myocardial infarction [Count of Participants; unit: Participants] | 7 | 3 | 10
Prior percutaneous coronary intervention [Count of Participants; unit: Participants] | 13 | 14 | 27
Prior coronary artery bypass graft surgery [Count of Participants; unit: Participants] | 0 | 0 | 0
CCS angina grade III or IV [Count of Participants; unit: Participants] — Canadian Cardiovascular Society grading of angina pectoris - Grade I - Ordinary physical activity does not cause angina. Grade II - Slight limitation of ordinary activity. Grade III - Marked limitation of ordinary physical activity. Grade IV - Inability to carry on any physical activity without discomfort, anginal syndrome may be present at rest
  Participants | 14 | 13 | 27
Body mass index, [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (4.6) | 30.2 (7.2) | 29.6 (6.0)
Multivessel disease [Count of Participants; unit: Participants] | 21 | 17 | 38
Bifurcation location [Count of Participants; unit: Participants] — LAD/Diagonal - left anterior descending artery LCX/OM - left circumflex coronary artery/obtuse marginal
  Participants
    LAD/Diagonal | 33 | 36 | 69
    LCX/OM | 2 | 0 | 2
Calcification [Count of Participants; unit: Participants]
  Moderate | 25 | 27 | 52
  Severe | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Side Branch Compromise
Description: Number of participants with Side Branch (SB) compromise which is defined as SB DS > 70%, or dissection or TIMI < 3
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy | CBA/PTCA
Number analyzed (Participants) | 35 | 36
Participants | 7 | 9

2. Secondary Outcome: Number of Participants With SB Dissection
Description: Number of participants with SB dissection
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy | CBA/PTCA
Number analyzed (Participants) | 35 | 36
Participants | 1 | 0

3. Secondary Outcome: Number of Participants With TIMI < 3
Description: Number of participants with TIMI flow grade < 3
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy | CBA/PTCA
Number analyzed (Participants) | 35 | 36
Participants | 3 | 5

4. Secondary Outcome: Number of Participants With SB DS >70%
Description: Number of participants with Side Branch Diameter Stenosis (DS) > 70%
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy | CBA/PTCA
Number analyzed (Participants) | 35 | 36
Participants | 2 | 4

5. Secondary Outcome: Number of Participants With FFR Device Success
Description: Number of Participants with successfully deliver Fractional Flow Reserve (FFR) wire to desired SB distal segment
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy | CBA/PTCA
Number analyzed (Participants) | 35 | 36
Participants | 28 | 27

6. Secondary Outcome: Number of Patients With FFR Wire Workhorse Capability
Description: FFR Wire Workhorse Capability - Number of patients in which FFR wire was able to serve as rail to deliver additional interventional devices to target SB lesion
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rotational Atherectomy | CBA/PTCA
Number analyzed (Participants) | 35 | 36
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Day
Arm/Group | Rotational Atherectomy | CBA/PTCA
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 3/35 | 1/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotational Atherectomy (N=35) | CBA/PTCA (N=36)
Chest Pain (Cardiac disorders) | 0 | 1
Transient sidebranch closing (Cardiac disorders) | 0 | 1 — requiring stenting
LM dissection with contrast injecting (Surgical and medical procedures) | 1 | 0 — surgical and medical procedures as organ system? or cardiac as organ system?
Right CFA access side bleeding (Surgical and medical procedures) | 1 | 0
Dissection Minor (Cardiac disorders) | 1 | 0
Side branch closure (Cardiac disorders) | 1 | 0 — symptomatic EKG changes
Staged PCI pf p:CS-OM1 (Cardiac disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03115580/Prot_SAP_000.pdf